CLINICAL TRIAL: NCT00456547
Title: Coagulation Factor Changes Associated With Postpartum Hysterectomies
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Other Study IDs: 0524-020
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Obstetric Labor Complications; Hemorrhage; Complications; Cesarean Section
Keywords: Cesarean hysterectomy; Postpartum hemorrhage; Coagulation
MeSH Terms: conditions — Obstetric Labor Complications; Hemorrhage; Postpartum Hemorrhage; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Postpartum hysterectomy: Women that require postpartum hysterectomy for post-delivery bleeding.
  Interventions: Procedure: Blood Draw
- Cesarean delivery case controls: Women that deliver by cesarean that presented with risk factors for bleeding but did not require post delivery hysterectomy
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Blood was obtained for coagulation studies at 2 hours following hysterectomy or cesarean delivery.
  Other Names: postpartum coagulation disorder

SUMMARY:
The purpose of this study is to examine components of the coagulation system in women undergoing postpartum hysterectomy and to compare laboratory parameters of coagulation in these women to women at increased risk for a postpartum hysterectomy, but who do not have postpartum hemorrhage and a postpartum hysterectomy. During normal pregnancy, the hemostatic balance tips toward hypercoagulation. Non-obstetric surgical blood loss is associated with increased coagulation activity. We have observed that women undergoing a postpartum hysterectomy become hypocoagulable secondary to a consumptive coagulopathy and/or excessive fibrinolysis. This coagulopathy may lead to the administration of multiple blood products. Worldwide, postpartum hemorrhage is a leading cause of maternal death. Plasma levels of tissue plasminogen activator, urokinase plasminogen activator and their inhibitors increase during pregnancy. During labor and delivery activation of coagulation occurs with consumption of platelets, coagulation factors and inhibitors. Obstetric complications during delivery can excessively activate the coagulation system and disseminated intravascular coagulation may ensue. Current treatment for postpartum coagulopathy is non-specific and primarily consists of replacing blood components. If specific causes or markers of abnormal coagulation can be identified in women at risk, then it might be possible to target (with specific medications) specific abnormalities early in the process and decrease hemorrhage and the need for blood transfusions.

DETAILED DESCRIPTION:
All women scheduled for a Cesarean-hysterectomy will be asked to enroll in the study, as well as the women with the following diagnoses, which puts them at increased risk for Cesarean hysterectomy: placenta previa, placenta accreta, vaginal trial of labor after a previous Cesarean delivery.

Written, informed consent will be obtained from all subjects. A blood sample will be obtained shortly after admission to the hospital. In women who go on to have a hysterectomy, blood samples will be obtained at predefined time periods (at time of decision to perform hysterectomy, with every clinically indicated blood draw for coagulation tests, 2 hours after delivery. The next patient at risk of Cesarean hysterectomy, but who does not go on to have a hysterectomy, will serve as a cohort control. Blood samples will be drawn at 2 hours after delivery for coagulation testing. Baseline samples from all other study subjects will be discarded and no further blood work will be obtained. The primary outcome will be the the level of fibrinogen at 2 hours following delivery as a marker of consumptive coagulopathy.

Every patient at risk for hemorrhage has at least one peripheral intravenous cannula inserted upon admission to the Labor & Delivery Unit. A 2nd IV cannula is almost always placed, usually when the decision is made to proceed with a Cesarean delivery. All study subjects will have a 2nd IV cannula placed for drawing blood for study coagulation tests, and any other clinically indicated blood tests. The cannula will be connected to a stopcock with a "heparin lock" (cannula and stopcock are flushed with saline between aspirations) and left in place for 48 hours after delivery.

ELIGIBILITY:
Inclusion Criteria:

* All women scheduled for a Cesarean-hysterectomy will be asked to enroll in the study, as well as the women with the following diagnoses, that puts them at increased risk for Cesarean hysterectomy: placenta previa, placenta accreta, vaginal trial of labor after previous Cesarean delivery.

Exclusion Criteria:

* Anyone who does not fit the above criteria.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2003-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Tuman KJ, Spiess BD, McCarthy RJ, Ivankovich AD. Effects of progressive blood loss on coagulation as measured by thrombelastography. Anesth Analg. 1987 Sep;66(9):856-63. PMID 3619091
- [Background] Hellgren M. Hemostasis during normal pregnancy and puerperium. Semin Thromb Hemost. 2003 Apr;29(2):125-30. doi: 10.1055/s-2003-38897. PMID 12709915
- [Background] Lanir N, Aharon A, Brenner B. Procoagulant and anticoagulant mechanisms in human placenta. Semin Thromb Hemost. 2003 Apr;29(2):175-84. doi: 10.1055/s-2003-38833. PMID 12709921
- [Background] Saftlas AF, Olson DR, Atrash HK, Rochat R, Rowley D. National trends in the incidence of abruptio placentae, 1979-1987. Obstet Gynecol. 1991 Dec;78(6):1081-6. PMID 1945212

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Postpartum Hysterectomy | Cesarean Delivery Case Controls
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postpartum Hysterectomy | Cesarean Delivery Case Controls | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Fibrinogen Level at 2 Hours After Delivery
Description: Fibrinogen level decrease is a marker of consumptive coagulation which is is a pathological activation of coagulation (blood clotting) mechanisms that happens in response to a variety of diseases or stimulus. We hypothesized that women with excessive bleeding following delivery who require a hysterectomy are more likely to exhibit lower levels of fibrinogen and a consumptive coagulopathy than women following cesarean delivery who do not bleed.
Time Frame: 2 hours after delivery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Postpartum Hysterectomy | Cesarean Delivery Case Controls
Number analyzed (Participants) | 12 | 12
mg/dL | 186 (80) | 418 (126)
Statistical Analysis 1: Comparison: Postpartum Hysterectomy vs Cesarean Delivery Case Controls; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Adjusted for 12 comparisons

2. Secondary Outcome: Platelet Counts at 2 Hours After Delivery
Description: Platelets are decreased in subjects with consumptive coagulopathies which is a pathological activation of coagulation (blood clotting) mechanisms that happens in response to a variety of diseases. We hypothesized that women who require hysterectomy for postpartum bleeding are more likely to have decreased platelet counts than matched controls that underwent cesarean delivery.
Time Frame: 2 hours after delivery
Measure: Mean (Standard Deviation); unit: platelets (*1000 per liter)
Arm/Group | Postpartum Hysterectomy | Cesarean Delivery Case Controls
Number analyzed (Participants) | 12 | 12
platelets (*1000 per liter) | 124 (30) | 179 (51)
Statistical Analysis 1: Comparison: Postpartum Hysterectomy vs Cesarean Delivery Case Controls; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Corrected for 12 comparisons

3. Secondary Outcome: Plasminogen Levels 2 Hours After Delivery
Description: Plasminogen is converted to plasmin when the coagulation system is activated. We hypothesized that plasminogen should be decrease more in women with continued bleeding following delivery requiring hysterectomy will demonstrated a greater decrease in plasminogen than following cesarean delivery.
Time Frame: 2 hours after delivery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Postpartum Hysterectomy | Cesarean Delivery Case Controls
Number analyzed (Participants) | 12 | 12
mg/dL | 66 (22) | 108 (26)
Statistical Analysis 1: Comparison: Postpartum Hysterectomy vs Cesarean Delivery Case Controls; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Corrected for 12 comparisons

4. Secondary Outcome: Antithrombin III Levels at 2 Hours Post Delivery
Description: Antithrombin III is a glycoprotein and is the major inhibitor of thrombin and other activated clotting factors, including factors IX, X, XI, and XII, the cofactor through which heparin exerts its effect. We hypothesized that women with continued bleed following delivery and require a hysterectomy will demonstrate a greater reduction in antithrombin III that women undergoing cesarean delivery.
Time Frame: 2 hours after delivery
Measure: Mean (Standard Deviation); unit: percentage of normal antithrombin III
Arm/Group | Postpartum Hysterectomy | Cesarean Delivery Case Controls
Number analyzed (Participants) | 12 | 12
percentage of normal antithrombin III | 51 (22) | 89 (18)
Statistical Analysis 1: Comparison: Postpartum Hysterectomy vs Cesarean Delivery Case Controls; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — Corrected for 12 comparisons

ADVERSE EVENTS:
Description: Adverse events were not collected as part of this study. The study protocol was a blood drawn and no additional follow-up was performed.
Arm/Group | Postpartum Hysterectomy | Cesarean Delivery Case Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes